CLINICAL TRIAL: NCT03186456
Title: Study the Safety and Efficacy of Human Umbilical Cord-derived Mesenchymal Stem Cells in the Treatment of Acute Cerebral Infarction
Brief Title: The Safety and Efficacy of Human Umbilical Cord Mesenchymal Stem Cells (19#iSCLife®-ACI) in the Treatment of Acute Cerebral Infarction
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Others
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCLnow-IMIMH-02
Record Dates: First submitted 2017-06-06; First posted 2017-06-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Infarction
Keywords: acute cerebral infarction; umbilical cord mesenchymal stem cells
MeSH Terms: conditions — Cerebral Infarction | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Aspirin Tablet, 100mg/d; Allogeneic umbilical cord mesenchymal stem cells, 0.5-1*10^6/kg
  Interventions: Biological: Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#); Drug: Aspirin Tablet
- Group 2 (Placebo Comparator): Aspirin Tablet, 100mg/d; Placebo
  Interventions: Drug: Aspirin Tablet

INTERVENTIONS:
Biological: Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#) — Allogeneic umbilical cord mesenchymal stem cells will transfusion into by forearm intravenous transplantation, 0.5 - 1 *10^6/kg. once a month, total 3 times.
  Arms: Group 1
Drug: Aspirin Tablet — Drug: Aspirin Tablet, 100 mg/d

SUMMARY:
The purposes of the study is to determine the safety and efficacy of treating acute ischemic stroke patients with human umbilical cord mesenchymal stem cells (hUC-MSC).

DETAILED DESCRIPTION:
This is a randomized, double-blind, paralleled study. 40 patients will be separated into two groups, and receive basic treatment (Aspirin Tablet). Patients in experimental group will receive hUC-MSC once a month, total 3 times. After the treatment, investigator will have follow-up visit for 6 months, evaluate the security and efficacy of hUC-MSC.

ELIGIBILITY:
Inclusion Criteria:

* Patient within 2 weeks onset of symptoms.
* Symptoms and signs of clinically definite acute cerebral infarction patients.
* CT/MRI prove the Oxfordshire Community Stroke Project (OCSP) as Total Anterior circulation infarct (TACI), Partial Anterior circulation infarct (PACI), Posterior Anterior circulation infarct (POCI), or obvious neurological deficit lacunar infarction patient.
* Signed informed consent after understanding all possible benefits and harm.

Exclusion Criteria:

* allergic to basic drug
* with progressive stroke, transient ischemia attach, cerebral infarction with posterior cerebral hemorrhage, and cerebral arteritis.
* tumor, injury, and parasites caused cerebral embolism
* rheumatic heart disease, coronary heart disease, and other atrial fibrillation combined heart disease caused cerebral embolism
* subject is processing thrombolytic therapy
* subject is pregnancy and of childbearing potential or breast feeding
* participate in any other clinical trial in last 3 months
* bleeding tendency patient; severe bleeding tendency in last 3 month
* with gastric duodenal ulcer
* participants with severe liver and kidney, hematopoietic, and metabolic diseases; Or with liver and kidney function examination abnormal
* participants are intolerance with Aspirin Enteric-coated Tablets, or need other antiplatelet drugs
* participants: alcoholism, drug addicted, or other situations may complicated the results
* under other therapy that possibly influence MSC security or efficacy
* investigator supposes not suitable to participate this clinical trail

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment related-adverse events counting | 26 weeks
  patients will be monitored for any adverse events resulting from the treatment of Human Umbilical Cord Mesenchymal Stem Cells

SECONDARY OUTCOMES:
Modified Rankin Scale | 26 weeks
  After the first time transplantation, follow-up visit for 26 weeks. Based on Modified Rankin Scale, counting the percentage of different symptom changes to evaluate MSC efficacy:
  * the percentage of participants run from 0-1, no symptom or no significant disability.
  * the percentage of participants run from 0-2, no symptom or slight disability.
  * the percentage of participants decline 2 scales compare to baseline.
  * the percentage of participants decline 1 scale compares to baseline.
Barthel activities of daily living (ADL) Index | 26 weeks
  Based on Activity of Daily Living Scale (ADL) to counting the percentage of patients in following condition:
  * the percentage of patients with score > 75
  * the decline of Barthel ADL Index range compares to baseline. Evaluate the efficacy of MSCs treatment
NIH stroke scale (NIHSS) | 26 weeks
  According to NIHSS changes after the treatment, evaluate MSCs efficacy by counting the percentage of patients in following condition:
  * the percentage of patients with score 0-1;
  * the percentage of patients with score declined 7 compare to baseline;
  * the percentage of patients with score declined 50% compare to baseline;
  * the declined ranges compare to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Temuqile, Study Director — Inner Mongolia International Mongolian Hospital; Lei Guo, Dr., Study Chair — China-Japan Union Hospital, Jilin University
Locations (1):
- Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No